CLINICAL TRIAL: NCT03326362
Title: Effects of Strength Training Upon Biomechanical, Morphological and Inflammatory Parameters of Chronic Low Back Pain Patients
Brief Title: Effects of Strength Training in Chronic Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Juliana Pennone, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Juliana Pennone
Record Dates: First submitted 2017-10-01; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; strength training; biomechanics; inflammatory biomarkers
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity resistance training (HIRT) (Experimental): 12 weeks of two weekly training sessions, with at least 48 hours of interval between sessions. The HIRT performed the squat, deadlift and lunge exercises, as these exercises induce high core muscles activity. HIRT started with two weeks of low intensity exercises emphasizing the activation of core muscles (pelvic elevation with feet on the floor, "superman", static supine bridge on bosu), and the technique of the selected resistance exercises (e.g. squat, deadlift, and lunges). Participants performed 3 sets of 10 repetitions per exercise. In the third and forth weeks, participants performed the exercises from the previous weeks and also static unipedal forward flexion on bosu and dynamic unipedal forward flexion and the main exercises with a load corresponding to (50% of the 1 RM load (Brzycki, 1993).
  From the 5th to the 12th week, participants performed only the selected resistance exercises with progressive higher intensities (from 12RM to 8RM).
  Interventions: Other: Resistance training
- Low intensity resistance training (LIRT) (Active Comparator): 12 weeks of two weekly training sessions, with at least 48 hours of interval between sessions.The LIRT group performed very low intensity and volume exercises (i.e. 1 set per exercise). Exercises started with participants lying on a firm surface, with the back supported, knees bent and feet flat on the floor. Then, participants performed the following exercises: 1) inhaling and exhaling and then isometrically contract in gluteal and abdominal muscles for 20 seconds and relax; 2) raising the head, lifting the chin and shoulders toward the chest for 20 seconds and relax; 3) raising one knee towards the chest and raising the head and shoulders likewise in the second exercise for 20s, relaxing, and changing the leg.; 4) raising both knees towards the chest in the same time that raise the head and shoulder off the floor during 20 seconds and relax.
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — Comparison between high and low intensities trainings described in arms

SUMMARY:
Although it is known that chronic low back pain (CLBP) have a multifactorial etiology, the investigations about it are mostly specific to each investigation area, making difficult to understand this complex condition. The purpose of the study was to investigate CLBP from a multidisciplinary approach, analyzing biomechanical, morphological and inflammatory parameters aiming to compare the influence of two strength training protocols, one of low intensity and low volume (LIT) and one of high intensity and high volume (HIT). In both experiments, pain intensity and level of functional disability were analyzed (by analogue scale of pain and Oswestry Index), Ground Reaction Forces (GRF - AMTI BP600900 - 2000 force plate), kinematics of lower limbs (Inertial Sensors by Noraxon) and electromyography of the rectus abdominis, external oblique, lumbar multifidus, medial gluteus, vastus lateralis and biceps femoris muscles (TelemyoDTS) during gait and sit-to-stand, inflammatory cytokines by Multiplex in blood samples and cross-sectional area (CSA) of the lumbar multifidus by ultrasound imaging.

DETAILED DESCRIPTION:
The subjects with CLBP were randomly assigned to two groups: the high intensity resistance training (HIRT) group and the low intensity resistance training (LIRT) groups.

All of the participants were informed of the purposes and procedures involved in the study and signed an informed consent form before participation. The experimental protocol was approved by the Institutional Review Board.

The intervention for both groups consisted of 12 weeks of two weekly training sessions, with at least 48 hours of interval between sessions. The HIRT performed the squat, deadlift and lunge exercises, as these exercises induce high core muscles activity. HIRT started with two weeks of low intensity exercises emphasizing the activation of core muscles (pelvic elevation with feet on the floor, "superman", static supine bridge on bosu), and the technique of the selected resistance exercises (e.g. squat, deadlift, and lunges). Participants performed 3 sets of 10 repetitions per exercise. In the third and forth weeks, participants performed the exercises from the previous weeks and also static unipedal forward flexion on bosu and dynamic unipedal forward flexion and the main exercises with a load corresponding to (50% of the 1 RM load (Brzycki, 1993).This formula is applied in a test that the subject is encouraged to perform the maximal number of repetitions possible with a predetermined load. The chosen load must allow the subject to achieve a maximum of ten repetitions, which guarantee a good RM prediction. The weight lifted and repetitions performed are applied in the equation to calculate the 1 RM estimation.

From the 5th to the 12th week, participants performed only the selected resistance exercises (squat, deadlift and lundge) with progressive higher intensities (from 12RM to 8RM). A 3-min rest interval was allowed between sets and exercises.

The LIRT group performed very low intensity and volume exercises (i.e. 1 set per exercise). Exercises started with participants lying on a firm surface, with the back supported, knees bent and feet flat on the floor. Then, participants performed the following exercises: 1) inhaling and exhaling and then isometrically contract in gluteal and abdominal muscles for 20 seconds and relax; 2) raising the head, lifting the chin and shoulders toward the chest for 20 seconds and relax; 3) raising one knee towards the chest and raising the head and shoulders likewise in the second exercise for 20s, relaxing, and changing the leg.; 4) raising both knees towards the chest in the same time that raise the head and shoulder off the floor during 20 seconds and relax.

ELIGIBILITY:
Inclusion Criteria:

* Being ≥18 years old
* Present low back or lumbo-sacral pain and function restriction (i.e. >15% in the Oswestry Questionnaire) for 12 weeks or longer
* Do not present any functional anatomical-abnormalities, neuromuscular joint diseases and acute symptoms of pain
* Recent participation in an exercise program (at least 12 weeks)
* Pregnancy or diseases that can directly impact systemic inflammation (i.e: cancer, diabetes, hypertension)

Exclusion Criteria:

• Minimum adherence to the training protocol, defined as performing at least 75% of the training sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Electromyographic activity of lower limb muscles during walking and sit-to-stand. | 12 weeks
  Electromyographic signal (1500 Hz) will be obtained from rectus abdominis, left and right external oblique, left and right lumbar multifidus, gluteus medius of the dominant limb, biceps femoris of the dominant limb, and vastus lateralis of the dominant limb using a wireless device (TeleMyoDTS,,Noraxon,CITY, USA). The location of the electrodes followed the SENIAM project database. Before electrode placement, skin sites will be shaved and abraded to remove hair and dead skin. Bipolar active surface electrodes (Meditrace 200, Kendal, silver; recording diameter = 1 mm; inter-electrode distance = 1 cm) were used. Electromyographic signal will be filtered using a band pass fourth order Butterworth filter with cut off frequency of 20 Hz and 450Hz.EMG data will be normalized by 200ms RMS peak .
Kinematic data for the lower limbs during walking and sit-to-stand | 12 weeks
  Seven inertial sensors (9DOF - Myomotion Inertial designed by Noraxon) will be placed on the pelvis and bilaterally in thigh, shank and foot. Sensors will be used to obtain three-dimensional orientation of the lower limbs in relation to pelvis and relative lower limb joints angles. Ankle dorsiflexion, knee extension and hip flexion were presented as a positive angles. Kinematic data will be sampled at 100 Hz and low-pass filtered at 6 Hz (fourth-order, zero-lag, Butterworth).
Kinetic data for the lower limbs during walking and sit-to-stand | 12 weeks
  Vertical ground reaction force (GFR) data will be obtained using either one (i.e. sit-to-stand) or two (i.e walking) strain gauge force plates(AMTI BP600900 - 2000;Watertown, EUA).GFR data will be sampled at 200 Hz and low-pass filtered at 50 Hz (fourth-order, zero-lag, Butterworth), and normalized by bodyweight. Sit-to-stand GFR parameters will be: peak vertical force, time to peak vertical force, and load rate both for stand up phase and sit down phases. Selected walking kinematics parameters will be first and second vertical peak force, time to first and second vertical peaks, load rate, total impulse, maximal deflection (i.e. minimum force value between the peaks) and time to maximal deflection.
Inflammatory Parameters | 12 weeks
  Blood samples (10 ml) will be obtained from the antecubital vein. After collection, the blood will be centrifuged at 3000 rpm for 15 min at 4° degrees. Plasma and serum will be storage in plastic microtubes at -80° degrees for posterior analysis of cytokines production of each participant by a qualified professional.
  The Multiplex Analysis of Sample Protein Content will be performed: each 10 ml of collected blood sample will be incubated with the mixture of Megaplex microspheres and covered with the specific antibodies for 2 h. The detection of target antigens bounded to the microspheres will be performed with a mixture of biotinylated capture antibodies after incubation for 1 h followed by incubation with streptavidin labeled with phycoerithrin for 30 min. The microspheres will be then analyzed with the phycoerithrinMagpix® instrument (Life Technologies, Grand Island, NY, USA). Citokines concentration will be normalized to total protein concentration.
Cross sectional area of lumbar multifidus | 12 weeks
  Lumbar multifidus ultrasound images will be obtained (transverse orientation at L4 in both sides of the spine with the subjects in prone lying position) using a B-mode ultrasound with a 7.5-MHz linear-array probe (SonoAce R3, Samsung-Medison, Gangwon-do, South Korea).The multifidus location will be determined by palpation of the spinous process of L5 and L4. L5 is deep, small and blunted bony point lying at the center of the lumbo-sacraldepression, on progression in a cranial direction is the comparatively large spinous process of L4. Ultrasound images will be obtained with SonoaceR3 equipment and their measurements in Image Jsoftware. For each subjects will be calculated the mean of CSA of the right and left sides of the lumbar multifidus.

CONTACTS AND LOCATIONS:
Locations (1):
- Juliana Pennone, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blackburn SE, Portney LG. Electromyographic activity of back musculature during Williams' flexion exercises. Phys Ther. 1981 Jun;61(6):878-85. Bressel E1, Willardson JM, Thompson B, Fontana FE. Effect of instruction, surface stability, and load intensity on trunk muscle activity. J Electromyogr Kinesiol. 2009 Dec;19(6):e500-4. doi: 10.1016/j.jelekin.2008.10.006. Epub 2008 Dec 2. Carpes, FP, Reinehr, FB, and Mota, CB. Effects of a program for trunk strength and stability on pain, low back and pelvis kinematics, and body balance: A pilot study. J Bodyw Mov Ther 12: 22-30, 2008. Clark, D, Lambert, M, and Hunter, A. Muscle activation in the loaded free barbell squat: a brief review. J Strength Cond Res 26: 1169-1178, 2012 Escamilla, RF, Francisco, AC, Kayes, A V, Speer, KP, and Moorman III, CT. An electromyographic analysis of sumo and conventional style deadlifts. Med Sci Sport Exerc 34: 682-688, 2002. Kristensen, J and Franklyn-Miller A. Resistance training in musculoskeletal rehabilitation: a systematic review. Br J Sports Med 46: 719-726, 2012.